CLINICAL TRIAL: NCT07323628
Title: Patient Satisfaction After Prosthetic Rehabilitation of Mandibular Single Denture With Two Implants Using Different Attachments: A Randomized Clinical Trial
Brief Title: PEEK vs Metal Bar Attachments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sherif Aly Sadek (Other)
Responsible Party: Sponsor-Investigator, Sherif Aly Sadek, Associate Professor, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02-02-23
Record Dates: First submitted 2025-12-19; First posted 2026-01-07 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Edentulism in Lower Jaw
Keywords: Mandibular Implant Overdenture; PEEK Bar Attachment; Metal Bar Attachment; Patient Satisfaction; Edentulous Mandible; Marginal Bone Loss
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two parallel intervention arms. Each participant receives two mandibular implants followed by prosthetic rehabilitation using either a CAD/CAM fabricated PEEK bar attachment or a conventional metal bar attachment. Outcomes are assessed longitudinally over a 12-month follow-up period without crossover between groups.
Who Masked: Outcomes Assessor
Masking Description: Radiographic measurements of marginal bone loss and analysis of patient satisfaction scores are performed by an independent assessor who is blinded to group allocation. Participants and care providers are not blinded due to visible differences in bar materials and clinical procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEEK Bar Attachment Group (Experimental): Participants receive two dental implants placed in the mandibular canine regions. After osseointegration, the mandibular overdenture is retained using a CAD/CAM-fabricated polyetheretherketone (PEEK) bar attachment. Clinical and patient-reported outcomes are evaluated over a 12-month follow-up period.
  Interventions: Device: PEEK Bar Attachment
- Metal Bar Attachment Group (Active Comparator): Participants receive two dental implants placed in the mandibular canine regions. After osseointegration, the mandibular overdenture is retained using a conventional metal alloy bar attachment. Clinical and patient-reported outcomes are evaluated over a 12-month follow-up period.
  Interventions: Device: Metal Bar Attachment

INTERVENTIONS:
Device: PEEK Bar Attachment — A CAD/CAM-fabricated polyetheretherketone (PEEK) bar used to retain a mandibular implant-supported overdenture on two implants placed in the canine regions of the mandible.
  Arms: PEEK Bar Attachment Group
Device: Metal Bar Attachment — A conventional metal alloy bar used to retain a mandibular implant-supported overdenture on two implants placed in the canine regions of the mandible.
  Arms: Metal Bar Attachment Group

SUMMARY:
This study is being conducted to compare two types of bar attachments used to support lower dentures in patients who have lost all their lower teeth. Many people who wear a single lower denture experience problems with stability, chewing, and comfort. Placing two implants in the lower jaw and attaching the denture to a bar can greatly improve how well the denture stays in place.

Traditionally, these bars have been made from metal. While effective, metal bars can place higher stress on the bone around the implants, which may lead to more bone loss over time. A newer material, PEEK (polyetheretherketone), is lighter and has flexibility closer to natural bone. This may reduce stress on the implants and help protect the surrounding bone.

In this randomized clinical trial, patients are assigned to receive either a PEEK bar or a metal bar to retain their lower denture. All participants receive two implants placed in the canine region of the lower jaw, followed by a bar-retained overdenture after healing.

The study follows patients for 12 months and measures:

Marginal bone loss: how much bone is lost around each implant, assessed through radiographs.

Patient satisfaction: how comfortable and functional the denture feels, including stability, chewing, speech, hygiene, and overall handling.

Early results show that both types of bars support the denture well, but implants connected to PEEK bars tend to show less bone loss after several months compared to those connected to metal bars. Patient satisfaction is high in both groups, with slightly higher scores reported by patients using PEEK bars, although not significantly different.

This study may help dentists choose the best bar material to improve long-term implant health and denture comfort.

DETAILED DESCRIPTION:
This randomized, parallel-group clinical trial evaluates the clinical performance of CAD/CAM-fabricated PEEK bars compared with traditional metal bars for retaining mandibular single overdentures supported by two implants. The study includes 20 fully edentulous mandibular patients aged 40-70 years who report functional difficulties with a single lower denture.

All participants undergo placement of two dental implants in the mandibular canine regions using a two-stage surgical protocol. After osseointegration, patients are randomly assigned to one of two groups:

PEEK bar group: overdentures retained using a digitally designed and milled PEEK bar.

Metal bar group: overdentures retained using a conventional metal alloy bar.

The scientific rationale for evaluating PEEK is based on its lower elastic modulus, which may allow more favorable stress distribution to peri-implant bone compared with the higher stiffness of metal bars. This biomechanical difference may influence implant survival, marginal bone remodeling, and perceived comfort.

Clinical outcomes are assessed at insertion and at 3, 6, 9, and 12 months. Marginal bone loss is measured radiographically using standardized periapical images. Patient-reported satisfaction is captured using a validated Visual Analogue Scale across major functional domains.

The statistical approach uses Aligned Rank Transform ANOVA due to non-normal data distribution, with Tukey post-hoc testing for pairwise comparison.

This trial contributes new data on material selection for bar attachments in implant-retained mandibular overdentures. The findings suggest that PEEK bars may offer biomechanical advantages by reducing bone loss while maintaining patient satisfaction comparable to metal bars. Further long-term studies with larger sample sizes are recommended to validate these results and support broader clinical adoption.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 40 to 70 years
* Mandibular single complete denture with complaints of poor retention or stability
* Adequate bone volume in the mandibular canine regions to receive two dental implants without the need for bone grafting
* Good general health allowing dental implant surgery
* Willingness to participate and comply with study procedures and follow-up visits
* Signed written informed consent

Exclusion Criteria:

* Presence of uncontrolled systemic diseases (e.g., uncontrolled diabetes mellitus)
* History of head and neck radiotherapy
* Metabolic bone diseases or conditions affecting bone healing
* Current smokers or tobacco users
* Poor oral hygiene or inability to maintain oral hygiene
* Active oral infections or untreated periodontal disease
* Bruxism or severe parafunctional habits
* Previous implant placement in the mandible
* Pregnant or lactating women

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-05-05 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction With Mandibular Implant-Retained Overdentures | Baseline (at overdenture insertion), and at 3, 6, 9, and 12 months post-insertion
  Description: Patient satisfaction will be evaluated using a Visual Analogue Scale (VAS). Participants will rate comfort, chewing efficiency, denture stability, speech, hygiene, ease of handling, and overall satisfaction. Scores will be recorded on a numerical scale and compared between intervention groups over the follow-up period.

SECONDARY OUTCOMES:
Marginal Bone Loss Around Dental Implants | Baseline (at overdenture insertion), and at 3, 6, 9, and 12 months post-insertion
  Description: Marginal bone loss around the two mandibular implants will be assessed radiographically using standardized periapical radiographs. Measurements will be recorded as the vertical distance (in millimeters) from the implant shoulder to the first bone-to-implant contact on the mesial and distal aspects of each implant. Mean bone loss per implant will be calculated and compared between the PEEK bar and metal bar attachment groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Nahda University, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tada, S., Stegaroiu, R., Kitamura, E., Miyakawa, O., & Kusakari, H. (2003). Influence of implant design on stress around implants. Journal of Prosthetic Dentistry, 90(2), 164-170.
- [Background] Schwitalla A, Muller WD. PEEK dental implants: a review of the literature. J Oral Implantol. 2013 Dec;39(6):743-9. doi: 10.1563/AAID-JOI-D-11-00002. Epub 2011 Sep 9. PMID 21905892
- [Background] Skalak R. Biomechanical considerations in osseointegrated prostheses. J Prosthet Dent. 1983 Jun;49(6):843-8. doi: 10.1016/0022-3913(83)90361-x. PMID 6576140
- [Background] Feine JS, Carlsson GE, Awad MA, Chehade A, Duncan WJ, Gizani S, Head T, Lund JP, MacEntee M, Mericske-Stern R, Mojon P, Morais J, Naert I, Payne AG, Penrod J, Stoker GT Jr, Tawse-Smith A, Taylor TD, Thomason JM, Thomson WM, Wismeijer D. The McGill Consensus Statement on Overdentures. Montreal, Quebec, Canada. May 24-25, 2002. Int J Prosthodont. 2002 Jul-Aug;15(4):413-4. No abstract available. PMID 12170858
- [Background] Burns DR. Mandibular implant overdenture treatment: consensus and controversy. J Prosthodont. 2000 Mar;9(1):37-46. doi: 10.1111/j.1532-849x.2000.00037.x. PMID 11074027